CLINICAL TRIAL: NCT02581306
Title: Exercise-mediated Changes in Adipocyte Differentiation and Metabolic Function
Brief Title: Exercise Induced Changes in Fat Metabolism
Acronym: BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor, Movement Science and Director, Substrate Metabolism Laboratory, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00103937
Record Dates: First submitted 2015-10-13; First posted 2015-10-20 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise session (Other): All subjects will exercise for 1 hour at a moderate intensity. There are no different arms in this study
  Interventions: Other: Exercise session

INTERVENTIONS:
Other: Exercise session — There is no drug or device intervention in this study. Subjects will exercise at a moderate intensity for 60 minutes and a blood sample will be obtained before and after the exercise session

SUMMARY:
If eligible to participate in the research study after completing the physical screening procedures, participants will be asked to return to the Substrate Metabolism Laboratory on another occasion after a short fast (no food or beverages - besides water) for at least 6 hours. After participants arrive, participants will rest quietly for approximately 30 min. The investigators will then collect a blood sample from a vein in participants hand, or forearm. After obtaining a baseline blood sample, participants will exercise at a moderate intensity (on a treadmill or a stationary bike) for one hour. This one hour moderate exercise session will feel like a slow jog during which participants would be able to carry a conversation. In order for the investigators to measure energy expended and the amount of fat participants are burning during exercise, the investigators will periodically ask participants to breathe through a mouthpiece so the investigators can collect participants expired breath. After the exercise session the investigators will collect another blood sample from a vein in participants hand, or forearm.

DETAILED DESCRIPTION:
General study design

* Subjects who exercise regularly will be instructed to exercise exactly 3 days before the experimental trial, and then abstain from their exercise training program until after the experiment is complete.
* Subjects will arrive to the Substrate Metabolism Laboratory (1210 CCRB) after at least a 6h fast.
* After resting quietly in the laboratory for approximately 30min, Dr. Horowitz will collect a resting blood sample by venipuncture, as he has done in our other IRB approved protocols (e.g., HUM00029179). Briefly, Dr. Horowitz will wash his hands and put on gloves. The participant's skin will be disinfected at the venipuncture site with isopropyl alcohol. Single-use needles will be used for each participant and immediately discarded into a biohazard sharps container after use. After the blood draw, direct pressure will be applied to the site of needle insertion to avoid/reduce bruising and discomfort.
* Subjects will exercise (bike or treadmill) for 1h at a moderate exercise intensity (approximately 65% of their predicted VO2peak). This moderate exercise intensity has been used extensively by Dr. Horowitz's laboratory in previous exercise testing and training studies in both lean and obese individuals, and is well tolerated by both populations.

  * During the exercise session, subjects will wear a heart rate monitor to ensure participants are exercising at the correct exercise intensity.
  * Subjects will also use the mouthpiece and nose clip (described above) for ~5min at the beginning, middle, and end of exercise to verify they are exercising at approximately 65% of their predicted VO2peak.
  * A study team member will be present with the participant at all times during exercise to ensure the comfort and safety.
* Immediately after exercise another blood sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Body Mass Index: 20-35 kg/m2
* Women must have regularly occurring menses and must be premenopausal

Exclusion Criteria:

* Pregnant or lactating
* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05-11 (Actual); Study Completion 2016-05-11 (Actual)

PRIMARY OUTCOMES:
changes in plasma concentrations of epinephrine after a session of exercise | 1 day
  Plasma levels will be measured using appropriate commercially available assays.
changes in plasma concentrations of lactate after a session of exercise | 1 day
  Plasma levels will be measured using appropriate commercially available assays.
changes in plasma concentrations of fatty acids after a session of exercise | 1 day
  Plasma levels will be measured using appropriate commercially available assays.
changes in plasma concentrations of IL-6 after a session of exercise | 1 day
  Plasma levels will be measured using appropriate commercially available assays.
changes in plasma concentrations of irisin after a session of exercise | 1 day
  Plasma levels will be measured using appropriate commercially available assays.
changes in plasma concentrations of growth hormone after a session of exercise | 1 day
  Plasma levels will be measured using appropriate commercially available assays.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States